CLINICAL TRIAL: NCT01302808
Title: A Phase I/II Study of Erlotinib and Romidepsin in Advanced Non-Small Cell Lung Cancer
Brief Title: Romidepsin and Erlotinib Hydrochloride in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Celgene (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, David E Gerber, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 012011-004; CDR0000653093 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-01035 (Registry Identifier: CTRP (Clinical Trials Reporting System)); STU 012011-004 (Other: UTSW)
Record Dates: First submitted 2011-02-19; First posted 2011-02-24 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: recurrent non-small cell lung cancer; stage III B non-small cell lung cancer; stage IV non-small cell lung cancer; malignant pleural effusion; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Erlotinib Hydrochloride; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Erlotinib plus Romidepsin (8 mg/m^2)) (Experimental): Erlotinib 150 mg orally daily plus romidepsin IV days 8 mg/m^2 administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle.
  Interventions: Combination Product: Erlotinib plus Romidepsin (8 mg/m^2)
- Cohort 2 (Erlotinib plus Romidepsin (10 mg/m^2)) (Experimental): Erlotinib 150 mg orally daily plus romidepsin IV days 10 mg/m^2 administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle.
  Interventions: Combination Product: Erlotinib plus Romidepsin (10 mg/m^2)
- Cohort 3 (Erlotinib plus Romidepsin (10 mg/m^2)) + Antiemetic prophylaxis (Experimental): Erlotinib 150 mg orally daily plus romidepsin IV days 10 mg/m^2 with antiemetic prophylaxis administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle.
  Interventions: Combination Product: Erlotinib plus Romidepsin (10 mg/m^2) + Antiemetic prophylaxis
- Cohort 4 (Erlotinib plus Romidepsin (8 mg/m^2)) + Antiemetic prophylaxis (Experimental): Erlotinib 150 mg orally daily plus romidepsin IV days 8 mg/m^2 with antiemetic prophylaxis administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle.
  Interventions: Combination Product: (Erlotinib plus Romidepsin (8mg/m^2)) + Antiemetic prophylaxis

INTERVENTIONS:
Combination Product: Erlotinib plus Romidepsin (8 mg/m^2)
  Other Names: Istodax®
  Arms: Cohort 1 (Erlotinib plus Romidepsin (8 mg/m^2))
Combination Product: Erlotinib plus Romidepsin (10 mg/m^2)
  Other Names: Istodax®
  Arms: Cohort 2 (Erlotinib plus Romidepsin (10 mg/m^2))
Combination Product: Erlotinib plus Romidepsin (10 mg/m^2) + Antiemetic prophylaxis
  Arms: Cohort 3 (Erlotinib plus Romidepsin (10 mg/m^2)) + Antiemetic prophylaxis
Combination Product: (Erlotinib plus Romidepsin (8mg/m^2)) + Antiemetic prophylaxis
  Arms: Cohort 4 (Erlotinib plus Romidepsin (8 mg/m^2)) + Antiemetic prophylaxis

SUMMARY:
RATIONALE: Romidepsin and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of romidepsin when given together with erlotinib hydrochloride and to see how well they work in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To characterize the toxicity and determine the maximum-tolerated dose (MTD) of erlotinib hydrochloride plus romidepsin. (Phase I)
* To obtain preliminary data regarding efficacy, including response rate and progression-free survival. (Phase II)

Secondary

* To characterize the pharmacokinetic profile of romidepsin in combination with erlotinib hydrochloride.
* To evaluate the impact of erlotinib hydrochloride on the biologic activity of romidepsin by analyzing peripheral blood mononuclear cell (PBMC) histone acetylation status and histone acetylase activity. (Exploratory)
* To evaluate the effect of romidepsin and erlotinib hydrochloride on components of the EGFR (epidermal growth factor receptor)-signaling pathway in skin biopsies, particularly downstream mediators such as MAPK (mitogen-activated protein kinase). (Exploratory)

OUTLINE: This is a dose-escalation study of romidepsin followed by a phase II study.

Patients receive romidepsin IV on days 1, 8, and 15 and erlotinib hydrochloride orally (PO) once daily beginning on day 3 of course 1 and on days 1-28 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for pharmacokinetic studies. Additional samples of peripheral blood mononuclear cells and skin biopsies may be also collected for correlative studies.

After completion of study therapy, patients are followed up for 30 days.

PROJECTED ACCRUAL: A total of 39 patients (15 patients for phase I and 24 patients for phase II) will be accrued for this study.

ELIGIBILITY:
To be eligible for study participation, patients must fulfill all of the following criteria:

* Histologically confirmed locally advanced or metastatic (stage IIIB pleural effusion or stage IV) NSCLC;
* Age ≥ 18 years;
* Written informed consent;
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST);
* ECOG (Eastern Cooperative Oncology Group ) performance status 0 to 1;
* Serum potassium and magnesium greater than or equal to the lower limit of institutional normal range (electrolyte abnormalities may be corrected with supplementation to meet inclusion criteria);
* Negative urine or serum pregnancy test on females of childbearing potential;
* All women of childbearing potential must use an effective barrier method of contraception (an intrauterine contraceptive device [IUCD] or double barrier method using condoms or a diaphragm plus spermicide) during the treatment period and for at least 1 month thereafter. Male patients should use a barrier method of contraception during the treatment period and for at least 1 month thereafter. Hormonal methods of contraception such as the contraceptive pill or patch (particularly those containing ethinyl-estradiol) should be avoided due to a potential drug interaction (see Appendix D).
* Adequate bone marrow, liver, and renal function as evidenced by
* Hemoglobin ≥10 g/dL (transfusions and/or erythropoietin-stimulating agents are permitted)
* Absolute neutrophil count (ANC) ≥1.5 x 109 cells/L • Platelet count ≥100 x 109 cells/L
* Total bilirubin <1.5 x upper limit of normal (ULN)
* (Aspartate amino transferase) AST/SGOT(serum glutamic-oxaloacetic transaminase) and (amino alanine transferase) ALT/SGPT (serum glutamic-pyruvic transaminase) <2.0 x upper limit of normal (ULN) or <3.0 x ULN in the presence of demonstrable liver metastases
* Serum creatinine <2.0 x ULN
* Clinically stable brain metastases are permitted

Phase I study:

* Prior erlotinib therapy is permitted (with a 3-week washout period)
* Patients may have received prior anti-cancer therapy (with a 3-week washout period) or, at the discretion of the investigator, may be treatment-naïve

Phase II study:

* Patients must have received at least one and no more than two prior chemotherapy regimens for their advanced NSCLC
* Patients may not have received prior erlotinib

Patients are ineligible for entry if any of the following criteria are met:

* Chemotherapy for NSCLC within 3 weeks prior to study entry;
* Concomitant use of any other anti-cancer therapy;
* Concomitant use of any investigational agent;
* Use of any investigational agent within 4 weeks prior to study entry;
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome;
  * QTc interval (corrected QT interval) Myocardial infarction within 12 months prior to study entry;
  * Other significant ECG abnormalities including type II second-degree atrio ventricular (AV) block, third-degree AV block, or bradycardia (ventricular rate < 50 beats/min); o A history of coronary artery disease (CAD); eg, angina Canadian Class II-IV. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * An ECG recorded at screening showing significant ST depression (ST depression of ≥2 mm, measured from isoelectric line to the ST segment at a point 60 msec from the end of the QRS complex). If there is any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction < 40% by MUGA ( multiple gated acquisition) scan or <50% by echocardiogram and/or MRI;
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsades de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardiac defibrillator (AICD);
  * Hypertrophic cardiomyopathy or restrictive cardiomyopathy from prior treatment or other causes (if there is any doubt, see ejection fraction criteria above);
  * Uncontrolled hypertension (defined as blood pressure [BP] ≥160/95; or
  * Any cardiac arrhythmia requiring anti-arrhythmic medication;
* Serum potassium or serum magnesium below lower limit of institutional normal range (electrolyte abnormalities may be corrected with supplementation to meet inclusion criteria)
* Concomitant use of drugs that may cause a prolongation of the QTc interval .
* Concomitant use of CYP3A4 inhibitors
* Concomitant use of warfarin (due to a potential drug interaction);
* Clinically significant active infection (including known infection with human immunodeficiency virus [HIV], hepatitis B, or hepatitis C); l >480 milliseconds (msec);
* Major surgery or radiation within 2 weeks prior to study entry;
* Patients who are pregnant or breast-feeding;
* Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures;
* Prior exposure to romidepsin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E. Gerber, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis
Started | 3 | 7 | 4 | 3
Completed | 3 | 7 | 4 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis | Total
Number analyzed (Participants) | 3 | 7 | 4 | 3 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 3 | 1 | 10
  >=65 years | 2 | 2 | 1 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 1 | 8
  Male | 3 | 3 | 1 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 2 | 7 | 3 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities and Maximum Tolerated Dose (MTD)
Description: Dose limiting toxicities per Protocol definition using (CTCAE), Version 3.0
Time Frame: 12 months
Population: Only phase 1 data are reported here as the phase 2 component of the study was not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis
Number analyzed (Participants) | 3 | 7 | 4 | 3
Participants | 0 | 2 | 0 | 0
Statistical Analysis 1: Comparison: Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) vs Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) vs Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis vs Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis; Test type: Other; Maximum Tolerated Dose = 8

2. Secondary Outcome: Area Under the Concentration-time Curve (AUC0 t) of Romidepsin in Combination With Erlotinib
Description: AUC0 t was measured in the time interval from 0 to time (t) when the last blood sample is collected with a concentration above the limit of quantification.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose on Days 1 and 8
Population: After exhausting all means to obtain the data, we were only able to find data per dosage and not by cohort. Pharmacokinetic profile will not be affected by antiemetic prophylactic drug and therefore data were reported per dose.
  Only phase 1 data are reported here as the phase 2 component of the study was not performed.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- Erlotinib Plus Romidepsin Cohort 1 (8mg/m2) + Cohort 4 (Modified Prophylaxis @ 8 mg/m2): Erlotinib 150 mg orally daily plus romidepsin IV days 1, 8, 15 (dose escalated) every 28 days
  erlotinib
  romidepsin
- Cohort 2 (10mg/m2) +Cohort 3 ( Modified Prophylaxis @ 10 mg/m2): Erlotinib 150 mg orally daily plus romidepsin IV days 10 mg/m^2 administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle (cohort 2), with antiemetic prophylaxis administered as a 4-h intravenous infusion on days 1, 8, and 15 of a 28-day cycle (cohort 3).
Arm/Group | Erlotinib Plus Romidepsin Cohort 1 (8mg/m2) + Cohort 4 (Modified Prophylaxis @ 8 mg/m2) | Cohort 2 (10mg/m2) +Cohort 3 ( Modified Prophylaxis @ 10 mg/m2)
Number analyzed (Participants) | 6 | 11
ng*h/ml
  Dosing day / Day 1 | 1207.00 (529.01) | 2185.52 (717.14)
  Dosing day / Day 8 | 989.19 (244.65) | 1851.84 (726.62)

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/7 | 3/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 3/7 | 1/4 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) (N=3) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) (N=7) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis (N=4) | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis (N=3)
Acute Kidney Injury (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Erlotinib Plus Romidepsin (8 mg/m^2)) (N=3) | Cohort 2 (Erlotinib Plus Romidepsin (10 mg/m^2)) (N=7) | Cohort 3 (Erlotinib Plus Romidepsin (10 mg/m^2)) + Antiemetic Prophylaxis (N=4) | Cohort 4 (Erlotinib Plus Romidepsin (8 mg/m^2)) + Antiemetic Prophylaxis (N=3)
Nausea (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Vomiting (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Only phase 1 data are reported here as the maximum tolerated dose of romidepsin in combination with standard erlotinib 150 mg orally daily administration was 8 mg/m2. Therefore, it did not proceed to phase 2 (14 mg/m2 )

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes